CLINICAL TRIAL: NCT05081089
Title: A Four-arm Trial Comparing Artemether-lumefantrine With or Without Single-dose Primaquine and Sulphadoxine-pyrimethamine/Amodiaquine With or Without Single-dose Tafenoquine to Reduce P. Falciparum Transmission in Mali
Brief Title: Gametocytocidal and Transmission-blocking Efficacy of PQ in Combination With AL and TQ in Combination With SPAQ in Mali
Acronym: NECTAR3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 26257
Record Dates: First submitted 2021-09-13; First posted 2021-10-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2021-08

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination; Primaquine; fanasil, pyrimethamine drug combination; Amodiaquine; tafenoquine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This is a single blind randomised controlled trial. The treating physician and staff involved with assessing all laboratory outcomes of the study are blinded, but no placebo will be used. The study pharmacist will be unblinded and responsible for randomisation and treatment administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Artemether-lumefantrine (AL) (Active Comparator): Subjects will receive artemether-lumefantrine (AL) twice daily for 3 days.
  Interventions: Drug: Artemether-lumefantrine
- AL with 0.25mg/kg primaquine (PQ) (Experimental): Subjects will receive artemether-lumefantrine (AL) twice daily for 3 days and a single dose of 0.25mg/kg primaquine (PQ) on the first day of AL treatment.
  Interventions: Drug: Artemether-lumefantrine; Drug: Primaquine Phosphate
- Sulphadoxine-pyrimethamine with amodiaquine (SPAQ) (Active Comparator): Subjects will receive sulphadoxine-pyrimethamine with amodiaquine (SPAQ) once daily for 3 days.
  Interventions: Drug: Sulphadoxine-pyrimethamine with amodiaquine
- SPAQ with 1.66mg/kg tafenoquine (TQ) (Experimental): Subjects will receive sulphadoxine-pyrimethamine with amodiaquine (SPAQ) once daily for 3 days and a single dose of 1.66mg/kg tafenoquine (TQ) on the first day of SPAQ treatment.
  Interventions: Drug: Sulphadoxine-pyrimethamine with amodiaquine; Drug: Tafenoquine

INTERVENTIONS:
Drug: Artemether-lumefantrine — Tablets containing 20/80 mg artemether and 120/480 mg lumefantrine will be administered according to weight as per manufacturer guidelines.
  Other Names: Riamet
  Arms: AL with 0.25mg/kg primaquine (PQ); Artemether-lumefantrine (AL)
Drug: Primaquine Phosphate — The single dose of 0.25mg/kg PQ will be administered in an aqueous solution, according to a standard operating procedure (SOP) provided by the manufacturer.
  Other Names: Primaquine
  Arms: AL with 0.25mg/kg primaquine (PQ)
Drug: Sulphadoxine-pyrimethamine with amodiaquine — Sulfadoxine/pyrimethamine tablets contain 500mg sulfadoxine and 25mg pyrimethamine. Amodiaquine tablets contain 150mg amodiaquine (as hydrochloride). Tablets will be administered according to weight as per manufacturer guidelines.
  Other Names: Supyra
  Arms: SPAQ with 1.66mg/kg tafenoquine (TQ); Sulphadoxine-pyrimethamine with amodiaquine (SPAQ)
Drug: Tafenoquine — 100mg tafenoquine tablets are prepared into a 1mg/mL solution in water. Solution will be given according to weight as indicated per treatment arm in 5kg bands.
  Other Names: Arakoda
  Arms: SPAQ with 1.66mg/kg tafenoquine (TQ)

SUMMARY:
The purpose of this study is to compare the gametocytocidal and transmission reducing activity of artemether-lumefantrine (AL) with and without a single dose of 0.25mg/kg primaquine (PQ) and sulfadoxine-pyrimethamine with amodiaquine (SPAQ) with and without single dose of 1.66mg/kg tafenoquine (TQ). Outcome measures will include infectivity to mosquitoes at 2, 5 and 7 days after treatment, gametocyte density throughout follow-up, and safety measures including haemoglobin density and the frequency of adverse events.

DETAILED DESCRIPTION:
Full protocol available on request.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 10 years and ≤ 50 years
* G6PD-normal defined by Carestart rapid diagnostic test or the OSMMR2000 G6PD qualitative test
* Absence of symptomatic falciparum malaria, defined by fever on enrolment
* Presence of P. falciparum gametocytes on thick blood film at a density >16 gametocytes/μL (i.e. ≥ gametocytes recorded in the thick film against 500 white blood cells)
* Absence of other non-P. falciparum species on blood film
* Hemoglobin ≥ 10 g/dL
* Individuals weighing < = 80 kg
* No evidence of acute severe or chronic disease
* Written, informed consent

Exclusion Criteria:

* Women who are pregnant or lactating (tested at baseline). Urine and/or serum pregnancy testing (β-hCG) will be used.
* Detection of a non-P. falciparum species by microscopy
* Previous reaction to study drugs / known allergy to study drugs
* Signs of severe malaria, including hyperparasitemia (defined as asexual parasitemia > 100,000 parasites / μL)
* Signs of acute or chronic illness, including hepatitis
* The use of other medication (except for paracetamol and/or aspirin)
* Use of antimalarial drugs over the past 7 days (as reported by the participant)
* Clinically significant illness (intercurrent illness e.g., pneumonia, pre-existing condition e.g., renal disease, malignancy or conditions that may affect absorption of study medication e.g., severe diarrhea or any signs of malnutrition as defined clinically)
* Signs of hepatic injury (such as nausea and/or abdominal pain associated with jaundice) or known severe liver disease (i.e., decompensated cirrhosis, Child Pugh stage B or C)
* Signs, symptoms or known renal impairment
* Clinically significant abnormal laboratory values as determined by history, physical examination or routine blood chemistries and hematology values (laboratory guideline values for exclusion are hemoglobin < 10 g/dL, platelets < 50,000/μl, White Blood Cell count (WBC) < 2000/μl, serum creatinine >2.0mg/dL, or ALT or AST more than 3 times the upper limit of normal for age.
* Blood transfusion in the last 90 days.
* Consistent with the long half-life of tafenoquine, effective contraception should be continued for 5 half-lives (3 months) after the end of treatment.
* History of psychiatric disorders

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Change in mosquito infection rate assessed through membrane feeding assays (day 2 and day 7) | 3 days (days 0, 2 and 7): 7 day span
  Within person percent change (presented as percent reduction) in mosquito infection rate in infectious individuals from baseline (day 0, pre-treatment) to day 2 post treatment in the AL and AL-PQ arms, and day 7 post-treatment in the SPAQ and SPAQ-TQ.

SECONDARY OUTCOMES:
Change in mosquito infection rate assessed through membrane feeding assays (all timepoints) | 7 days (day 0, day 2, day 5, day 7, day 14, day 21, day 28): 28 day span
  Within person percent change (presented as percent reduction) in mosquito infection rate from baseline to all feeding time-points, with comparison within and between arms.
Mosquito infection rate assessed through membrane feeding assays | 7 days (day 0, day 2, day 5, day 7, day 14, day 21, day 28): 28 day span
  Mosquito infection rate at all feeding time-points, with comparison within treatment arms compared to baseline, and between arms.
Human infectivity to locally reared mosquitoes assessed through membrane feeding assays | 7 days (day 0, day 2, day 5, day 7, day 14, day 21, day 28): 28 day span
  Infectivity to mosquitoes at all feeding time-points, with comparison within treatment arms compared to baseline, and between arms.
Mosquito infection density assessed through membrane feeding assays | 7 days (day 0, day 2, day 5, day 7, day 14, day 21, day 28): 28 day span
  Oocyst intensity (in all/all infected mosquitoes) at all feeding time-points, with comparison within treatment arms compared to baseline, and between arms.
Gametocyte infectivity | 7 days (day 0, day 2, day 5, day 7, day 14, day 21, day 28): 28 day span
  Infectiousness to mosquitoes for a given gametocyte density (measured as mosquito infection rate/gametocyte) at all feeding time-points, with comparison within treatment arms compared to baseline, and between arms.
Asexual/sexual stage parasite prevalence | 7 days (day 0, day 2, day 5, day 7, day 14, day 21, day 28): 28 day span
  Male and female gametocyte prevalence at all time-points, determined by microscopy or molecular assays, with comparison within treatment arms compared to baseline, and between arms.
  Asexual and total parasite prevalence at all time-points, determined by microscopy or molecular assays, with comparison within treatment arms compared to baseline, and between arms.
Asexual/sexual stage parasite density | 7 days (day 0, day 2, day 5, day 7, day 14, day 21, day 28): 28 day span
  Male and female gametocyte density at all time-points, determined by microscopy or molecular assays, with comparison within treatment arms compared to baseline, and between arms.
  Asexual and total parasite density at all time-points, determined by microscopy or molecular assays, with comparison within treatment arms compared to baseline, and between arms.
Sexual stage parasite sex ratio | 7 days (day 0, day 2, day 5, day 7, day 14, day 21, day 28): 28 day span
  Male and female gametocyte sex ratio (proportion male) at all time-points, determined by microscopy or molecular assays, with comparison within treatment arms compared to baseline, and between arms.
Sexual stage parasite circulation time | 7 days (day 0, day 2, day 5, day 7, day 14, day 21, day 28): 28 day span
  Gametocyte circulation time (cumulative), determined by microscopy or molecular assays, compared within and between treatment arms.
Sexual stage parasite area under the curve (AUC) | 7 days (day 0, day 2, day 5, day 7, day 14, day 21, day 28): 28 day span
  Gametocyte area under the curve (cumulative), determined by microscopy or molecular assays, compared within and between treatment arms.
Haemoglobin density | 8 days (day 0, day 1, day 2, day 5, day 7, day 14, day 21, day 28): 28 day span
  Haemoglobin density (g/dL) at all time-points, with comparison within treatment arms compared to baseline, and between arms.
Change in haemoglobin density | 8 days (day 0, day 1, day 2, day 5, day 7, day 14, day 21, day 28): 28 day span
  Within person percent change (presented as percent reduction) in haemoglobin density (g/dL) from baseline to all time-points, with comparison within and between arms.
Methaemoglobin density | 8 days (day 0, day 1, day 2, day 5, day 7, day 14, day 21, day 28)
  Methaemoglobin density (g/dL) at all time-points, with comparison within treatment arms compared to baseline, and between arms.
Change in methaemoglobin density | 8 days (day 0, day 1, day 2, day 5, day 7, day 14, day 21, day 28): 28 day span
  Within person percent change (presented as percent reduction) in methaemoglobin density (g/dL) from baseline to all time-points, with comparison within and between arms.
Incidence of adverse events | 8 days (day 0, day 1, day 2, day 5, day 7, day 14, day 21, day 28): 28 day span
  The frequency and prevalence of adverse events (all AE's, treatment related AE's, and haematological AE's) observed up to and including day 2, 7, and 14 post-treatment, and at all timepoints.

OTHER OUTCOMES:
Parasite genomic and transcriptomic variation assessed in RNA | 7 days (day 0, day 2, day 5, day 7, day 14, day 21, day 28): 28 day span
  Parasite genotype and transcriptional analysis at baseline and at post-treatment timepoints.
The impact of plasma biomarkers on malaria transmission efficiency | 7 days (day 0, day 2, day 5, day 7, day 14, day 21, day 28): 28 day span
  Plasma biomarkers (antibodies and parasite protein) at baseline and at post-treatment timepoints.
Human genomic variation analysis and association with parasite measure | day 0
  Human genotype analysis at baseline (G6PD, CYP2D6, and HBB type)
ALT/AST/Creatine density | 8 days (day 0, day 1, day 2, day 5, day 7, day 14, day 21, day 28): 28 day span
  ALT/AST/Creatine density at all time-points with comparison within treatment arms compared to baseline, and between arms.

CONTACTS AND LOCATIONS:
Overall Officials: Alassane Dicko, Principal Investigator — Malaria Research and Training Centre, Mali
Locations (1):
- Malaria Research and Training Centre, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No
Anonymised individual participant data may be shared on a digital repository or upon reasonable request.

REFERENCES:
- [Derived] Mahamar A, Smit MJ, Sanogo K, Sinaba Y, Niambele SM, Sacko A, Dicko OM, Diallo M, Maguiraga SO, Sankare Y, Keita S, Samake S, Dembele A, Lanke K, Ter Heine R, Bradley J, Dicko Y, Traore SF, Drakeley C, Dicko A, Bousema T, Stone W. Artemether-lumefantrine with or without single-dose primaquine and sulfadoxine-pyrimethamine plus amodiaquine with or without single-dose tafenoquine to reduce Plasmodium falciparum transmission: a phase 2, single-blind, randomised clinical trial in Ouelessebougou, Mali. Lancet Microbe. 2024 Jul;5(7):633-644. doi: 10.1016/S2666-5247(24)00023-5. Epub 2024 May 2. PMID 38705163